CLINICAL TRIAL: NCT04344977
Title: A Pilot Study for Collection of Anti-SARS-CoV-2 Immune Plasma
Brief Title: Collection of Anti-SARS-CoV-2 Immune Plasma
Acronym: NIAID
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200081; 20-I-0081 (Other: NIHCC)
Record Dates: First submitted 2020-04-13; First posted 2020-04-14 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
Keywords: Coronavirus; COVID-19; IVIG; Convalescent plasma; Severe acute respiratory syndrome coronavirus 2
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Convalescent survivors of COVID-19: Convalescent survivors of COVID-19: history of COVID-19 like illness or positive test for SARS-CoV-2 and has the protocol-specified minimum anti-SARS-CoV-2 neutralizing antibody titer

SUMMARY:
Background:

The human disease caused by SARS-CoV-2 is called COVID-19. In most cases, COVID-19 is a mild to moderate respiratory illness. But it can also be more severe and even lead to death. There is no vaccine to prevent SARS-CoV-2 infection. There is also no therapy to treat COVID-19. Researchers want to collect plasma from adults who have recovered from COVID-19, which may help them develop treatments.

Objective:

To collect anti-SARS-CoV-2 immune plasma from adult volunteers who have recovered from COVID-19.

Eligibility:

Males and females ages 18 to 70 who have a history of COVID-19 like illness or positive test for SARS-CoV-2, and have a minimum level of SARS-CoV-2 antibodies as specified by the study.

Design:

This study consists of 2 parts: 1) screening for SARS-CoV-2 antibody titer and eligibility to donate plasma and 2) plasma collection by apheresis. Study sites may participate in 1 part alone (either screening or plasma collection only) or both parts (screening and plasma collection).

For screening part: Participants will be screened for their eligibility to join this research study with a medical history and physical exam. Their vital signs (blood pressure, heart rate, temperature, respiration rate) will be taken. Their weight and height will be recorded. They will give a blood sample for clinical laboratory tests of their general health and a research test for SARS-CoV-2 antibodies. They will discuss their history of COVID-19-like illness and any testing for SARS-CoV-2. They will be evaluated for their ability to donate plasma.

For plasma collection part: Subjects meeting criteria for plasma donation and found to have high neutralizing antibody titers and who plan to donate plasma under this part of the study will be scheduled for 1 (and up to 20) plasma collection sessions. These will occur no less than 7 days apart.

Prior to each donation, participants will have a brief physical exam and complete a donor history questionnaire. They will be asked about any current SARS-CoV-2 infection symptoms.

At each donation, plasma will be taken through a standard apheresis procedure. For this, blood will be withdrawn through a needle placed in the participant's arm vein. A machine will separate the plasma from the red cells. The red cells will be returned to the participant, either through the same needle or through a second needle in the other arm.

Participation may last up to 240 days.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is a respiratory disease caused by a novel coronavirus named severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and causes substantial morbidity and mortality. There is currently no vaccine to prevent infection with SARS-CoV-2 or therapeutic agent to treat COVID-19. The objective of this protocol is the identification of eligible donors and collection of anti-SARSCoV-2 immune plasma from convalescent survivors of COVID-19 illness.

Potential subjects will be screened for eligibility to participate in plasma donations and their blood measured for antibodies to SARS-CoV-2. Enrolled subjects will receive a baseline physical and laboratory examination. Subjects with high SARS-CoV-2 neutralizing antibody titers who meet standard blood bank criteria for plasma donation will then be scheduled for plasma collection sessions. Following testing of the collected plasma for potential pathogens, this plasma may be used and/or converted into an intravenous immunoglobulin (IVIG) preparation for further study.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Provide written informed consent before initiation of any study procedures.
2. Age greater than or equal to 18 years old and less than or equal to 70 years old.
3. Subjects must not be symptomatic, must be afebrile for ≥14 days, beyond 28 days of the resolution of their acute COVID-19 illness, and must enroll within 18 months of onset of illness, and must meet at least 1 of the following:

   * History suggestive of resolved COVID-19-like illness (e.g., prior fever, dry cough, and shortness of breath). OR
   * History of positive test for SARS-CoV-2 (either serologic or RT-PCR) OR
   * Documented anti-SARSCoV-2 neutralizing antibody titer of at least 1:80
4. Current anti-SARS-CoV-2 neutralizing antibody titer of at least 1:80
5. Females must have a negative anti-HLA screening test
6. Weight greater than or equal to110 pounds (50 kg)
7. Meets FDA-approved criteria per local blood collector for plasmapheresis for plasma donation
8. Adequate peripheral venous access for plasma donation (as judged by the examiner)
9. Willingness to have samples stored

EXCLUSION CRITERIA:

1. Any sign of active illness of any kind including COVID-19 illness (as judged by the investigator), including but not limited to:

   * Subjective or documented fever (greater than or equal to 38°C)
   * Dry cough
   * Shortness of breath
2. Participation in medical research that includes:

   * Protocols that are currently ongoing or will start during the duration of this study that require more than 100 mL of blood to be given in any 8-week period of time
   * Administration of any unlicensed drug within the last 1 month or during the duration of this study, per investigation discretion
   * Administration of any unlicensed vaccine within the last 12 months or during the duration of this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Convalescent survivors of COVID-19 will be recruited at sites around the US.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Identification of eligible donors and collection of anti-SARS-CoV-2 immune plasma | Screening, Days 120 or 240
  Donors screened and identified and anti-SARS-CoV-2 immune plasma collected

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Lundquist Institute for Biomedical Innovation at Harbor - UCLA Medical Center, Torrance, California
  - University of Miami Infectious Diseases Research Unit, Miami, Florida
  - Bloodworks Northwest, Seattle, Washington